CLINICAL TRIAL: NCT04139005
Title: Well-being and the Healthy Minds App Pilot (WHAP) Study
Brief Title: Well-being and the HM App Pilot (WHAP) Study
Acronym: WHAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-0893; A538900 (Other: UW Madison); SMPH/PSYCHIATRY/PSYCHIATRY (Other: UW Madison)
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2020-10

CONDITIONS: Well-being
MeSH Terms: interventions — Immunization Programs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Awareness-Connection (Experimental)
  Interventions: Behavioral: Awareness; Behavioral: Connection
- Awareness-Insight (Experimental)
  Interventions: Behavioral: Awareness; Behavioral: Insight
- Wait list (No Intervention)

INTERVENTIONS:
Behavioral: Awareness — The program foundation targets attention and awareness skills that are integral to many conceptions of mindfulness.
  Other Names: Healthy Minds Program
  Arms: Awareness-Connection; Awareness-Insight
Behavioral: Connection — The Connection module targets skills underlying social connection, which refers to the sense of having close and positively experienced relationships with others in the social world.
  Other Names: Healthy Minds Program
  Arms: Awareness-Connection
Behavioral: Insight — The Insight module targets skills underlying dynamic self-inquiry and experiential self-knowledge.
  Other Names: Healthy Minds Program
  Arms: Awareness-Insight

SUMMARY:
There is no single definition of well-being, but consensus exists that positive functioning beyond the absence of detrimental mental health symptoms is central. Building on related "eudaimonic" frameworks of psychological flourishing that identify qualities like environmental mastery, positive relations with others, and personal growth, this study targets brain-based skills that underlie the active cultivation of such qualities (e.g., regulating attention, empathic care, mental flexibility), and thus offers straightforward hypotheses about mechanisms of change.

The Healthy Minds Program (HMP) is designed to promote and protect psychological well-being through sustainable skills training. The program is grounded in constituents of psychological well-being identified in empirical literature. HMP provides core content, with instruction administered through a curriculum of high-quality guided practices. HMP is based on research on eudaimonic well-being (e.g., environmental mastery, purpose) and brain-based skills that underlie these qualities (e.g., regulation of attention, mental flexibility). HMP practices address 4 constituents of well-being: awareness, connection, insight, and purpose. This pilot focuses on awareness, connection, and insight.

ELIGIBILITY:
Inclusion Criteria:

* Between the age of 18-65

Exclusion Criteria:

* Individuals under 18 or over 65
* Significant meditation experience (as defined below):
* Meditation retreat experience (meditation retreat or yoga/body practice retreat with significant meditation component).
* Regular meditation practice weekly for over 1 year OR daily practice within the previous 6 months.
* Previous practice under the instruction of a meditation teacher, other than in the context of an introductory course.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Change in Depression symptoms as assessed by PROMIS Depression score | Baseline, 4-6 weeks, 10-12 weeks, 3 month follow-up, 6 month follow-up, 9 month follow-up
  Self-reported experience of depression symptoms over the past 7 days. Eight items are scored on a scale of 1-5 (1 = never experience, 5 = always experience).
Change in Anxiety symptoms as assessed by PROMIS Anxiety score | Baseline, 4-6 weeks, 10-12 weeks, 3 month follow-up, 6 month follow-up, 9 month follow-up
  Self-reported experience of anxiety symptoms over the past 7 days. Eight items are scored on a scale of 1-5 (1 = never experience, 5 = always experience).
Change in Perceived Stress Scale | Baseline, 4-6 weeks, 10-12 weeks, 3 month follow-up, 6 month follow-up, 9 month follow-up
  Self-reported stressful experiences over the past month. Fourteen items are scored on a scale of 0-4 (0 = never experience, 4 = very often experience).
Change in the Social Connectedness Scale score | Baseline, 4-6 weeks, 10-12 weeks, 3 month follow-up, 6 month follow-up, 9 month follow-up
  Self-reported feelings related to social connection. Twenty items are scored on a scale of 1-6 (1 = strongly disagree, 6 = strongly agree).
Change in Dispositional empathy as assessed by Interpersonal Reactivity Scale | Baseline, 4-6 weeks, 10-12 weeks, 3 month follow-up, 6 month follow-up, 9 month follow-up
  Self-reported thoughts and feelings related to empathy. Twenty-eight items are scored on a scale of A-E (A = does not describe me well, E = describes me very well).
Change in Compassion as assessed by Compassionate Love Scale | Baseline, 4-6 weeks, 10-12 weeks, 3 month follow-up, 6 month follow-up, 9 month follow-up
  Self-reported feelings of compassion for close others and humanity. Twenty-one items are scored on a scale of 1-7 (1 = not true at all of me, 7 = very true of me).
Change in Self-Reflection and Insight Scale score | Baseline, 4-6 weeks, 10-12 weeks, 3 month follow-up, 6 month follow-up, 9 month follow-up
  Self-reported thoughts of introspection and self-understanding. Twenty items are scored on a scale of 1-6 (1 = strongly disagree, 6 = strongly agree).
Change in repetitive negative thinking as assessed by Perseverative Thinking Questionnaire score | Baseline, 4-6 weeks, 10-12 weeks, 3 month follow-up, 6 month follow-up, 9 month follow-up
  Self-reported experiences with negative thoughts. Fifteen items are scored on a scale of 0-4 (0 = never, 4 = almost always).
Change in the Defusion as assessed by Drexel Defusion Scale | Baseline, 4-6 weeks, 10-12 weeks, 3 month follow-up, 6 month follow-up, 9 month follow-up
  Self-reported distancing from internal experiences during difficult hypothetical situations. Ten items are scored on a scale of 0-5 (0 = not at all, 5 = very much).

SECONDARY OUTCOMES:
App Usage as assessed by number of logins | up to 9 month follow-up
  Number of logins as tracked by the intervention app.
App Usage as assessed by minutes of practice each day | up to 9 month follow-up
  Minutes of practice as tracked by the intervention app.
Change in the Mindfulness (Five Factor Mindfulness Questionnaire) | Baseline, 4-6 weeks, 10-12 weeks, 3 month follow-up, 6 month follow-up, 9 month follow-up
  Self-reported mindfulness during typical daily experiences. Thirty-nine items are scored on a scale of 1-5 (0 = never or very rarely true, 5 = very often or always true).

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Rosenkranz, PhD, Principal Investigator — University of Wisconsin, Madison; Simon Goldberg, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Center for Healthy Minds, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Any collected data may be made anonymous and transmitted through shared folders, via email, by usb, or other avenues and made available upon request or shared publicly in an open science format.
  All identifiers (i.e., names, contact information, date of birth, visit dates) will be stripped to assure confidentiality of this data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data may be shared following analysis and publication or upon request.

REFERENCES:
- [Derived] Goldberg SB, Imhoff-Smith T, Bolt DM, Wilson-Mendenhall CD, Dahl CJ, Davidson RJ, Rosenkranz MA. Testing the Efficacy of a Multicomponent, Self-Guided, Smartphone-Based Meditation App: Three-Armed Randomized Controlled Trial. JMIR Ment Health. 2020 Nov 27;7(11):e23825. doi: 10.2196/23825. PMID 33245288